CLINICAL TRIAL: NCT01212965
Title: Pilot Clinical Trial to Estimate the Safety and Efficacy of Selenium in the Treatment of Complicated Lymphatic Malformations in Adolescents and Young Adults
Brief Title: Selenium in the Treatment of Complicated Lymphatic Malformations
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The investigators chose to terminate the study due to participant attrition. Of the limited data evaluable, none of the patients experienced adverse events.
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Michael Kelly, Principal Investigator, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10/93
Record Dates: First submitted 2010-09-24; First posted 2010-10-01 (Estimated); Last update posted 2013-04-23 (Estimated); Status verified 2013-04

CONDITIONS: Lymphatic Malformations
Keywords: Selenium; Lymphatic Malformations; Adolescents
MeSH Terms: conditions — Lymphatic Abnormalities | interventions — Selenium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Selenium — 400 μg once a day for 6 months by mouth
  Other Names: Selenase

SUMMARY:
The investigators propose a pilot trial to obtain preliminary information regarding the safety and response rate of patients with symptomatic lymphatic malformations treated with oral Selenium. Information obtained in this pilot trial will be used to plan future phase 2 clinical trials.

Hypotheses:

* Selenium will be safe and efficacious in the treatment of adolescents and young adults with symptomatic lymphatic malformations
* Disease response will correlate with serum levels of selenium and blood levels of antioxidants essential to selenium metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have clinical and radiographic features consistent with a lymphatic malformation (LM). Patients with combined venous lymphatic malformations (CVLM) will be included if the predominant componet is lymphatic based on MRI. Both macrocystic and microcystic LM will be eligible. Tissue biopsy is required to confirm the presence of an abnormal lymphatic malformation.
* All patients diagnosed with lymphatic malformations between 14 and 30 years of age will be eligible.
* Patients must have lymphatic malformations with potential to cause morbidity including one or more of the following: Lymphedema, Coagulopathy, Chronic Pain, Recurrent Cellulitis (> 1 episodes/year), Ulceration and/or bleeding, Impairment of organ function, Visceral and/or bone involvement, or Disfigurement.
* Patients receiving previous systemic therapy, surgical, debulking, or sclerotherapy will be eligible eight weeks following completion of therapy if they meet all inclusion criteria.
* All patients and/or their parents or legal guardians must sign a written informed consent. All institutional FDA requirements for human studies must be met.

Exclusion Criteria:

* Younger than 14 years of age or older than 30 years of age
* Life-threatening complications related to LM
* Patients with preexisting renal, hepatic, or thyroid disorders
* Patients receiving a daily multivitamin supplement or other natural products that include selenium
* Patients that have received previous selenium therapy will not be eligible
* Women who are pregnant or breastfeeding

Ages: 14 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2010-09; Primary Completion 2011-09 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Determine a preliminary rate to oral selenium in adolescents and young adults with symptomatic lymphatic malformations | pretreatment and at 6 months
  Disease will be assessed by volumetric MRI and patient quality of life assessments at 6 months of therapy and compared to pretreatment values.
Determine the safety of oral selenium in adolescents and young adults with symptomatic lymphatic malformations | throughout duration of study

SECONDARY OUTCOMES:
Correlate selenium drug levels, expression of selenoproteins and IL-20with outcome | throughout duration of study
  Whole blood will be drawn prior to therapy and at specific time intervals after initiating selenium. Serum concentrations of selenium, selenium-dependent tripeptide glutathione and IL-20 will be measured and correlated with outcome

CONTACTS AND LOCATIONS:
Overall Officials: Michael E Kelly, MD, PhD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Children's Hospital of Wisconsin, Milwaukee, Wisconsin, United States